CLINICAL TRIAL: NCT00108758
Title: Exploratory, Multi-centre, Randomised, Double-blind, Uncontrolled Trial Evaluating the Efficacy of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in Secondary Bleeding Prophylaxis in Congenital Haemophilia A or B Patients With Inhibitors
Brief Title: Efficacy of NovoSeven® in Bleeding Prophylaxis in Hemophilia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7HAEM-1505
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Africa, Asia, Europe, South America, and the United States of America (USA).

The purpose of this study is to evaluate the effectiveness of secondary prophylactic treatment with NovoSeven® in haemophilia A and B patients with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital haemophilia A or B with inhibitors development against FVIII or FIX, respectively

Exclusion Criteria:

* Prophylactic administration of any haemostatic drug within 3 last months prior to entering the trial.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Reduction of bleeds | During 3 months treatment period as compared to 3 months observation period

SECONDARY OUTCOMES:
Efficacy variables

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (35):
- United States (12):
  - Novo Nordisk Investigational Site, Berkeley, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas
- Novo Nordisk Investigational Site, Ciudad Autónoma de Bs. As., Argentina
- Brazil (5):
  - Novo Nordisk Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, Belo Horizonte
  - Novo Nordisk Investigational Site, Recife
  - Novo Nordisk Investigational Site, Ribeirão Preto
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- France (3):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Paris
- Novo Nordisk Investigational Site, Manila, Philippines
- Poland (3):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Warsaw
- Romania (2):
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Bucharest
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Johannesburg, Gauteng, South Africa
- Spain (3):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Capa-ISTANBUL

REFERENCES:
- [Result] Konkle BA, Ebbesen LS, Erhardtsen E, Bianco RP, Lissitchkov T, Rusen L, Serban MA. Randomized, prospective clinical trial of recombinant factor VIIa for secondary prophylaxis in hemophilia patients with inhibitors. J Thromb Haemost. 2007 Sep;5(9):1904-13. doi: 10.1111/j.1538-7836.2007.02663.x. PMID 17723130
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com